CLINICAL TRIAL: NCT06049576
Title: Combination Nivolumab and Ipilimumab With and Without Camu Camu in First Line Treatment of Metastatic Renal Cell Carcinoma
Brief Title: Nivolumab and Ipilimumab With and Without Camu Camu for the Treatment of Patients With Metastatic Renal Cell Carcinoma
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: met goal
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22457; NCI-2023-06703 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22457 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2023-09-07; First posted 2023-09-22 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Clear Cell Renal Cell Carcinoma; Sarcomatoid Renal Cell Carcinoma; Stage III Renal Cell Cancer AJCC v8; Stage IV Renal Cell Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Specimen Handling; Ipilimumab; CTLA-4 Antigen; Magnetic Resonance Spectroscopy; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (nivolumab and ipilimumab) (Active Comparator): Patients receive nivolumab IV over 30 minutes on day 1 and ipilimumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 3 weeks for cycles 1-4. Beginning cycle 5, patients receive nivolumab over 30 minutes on day 1 of each cycle. Cycles repeat every 4 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo blood and stool sample collection and undergo CT and/or bone scan and/or MRI on trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Biological: Ipilimumab; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab
- Arm 2 (nivolumab, ipilimumab, camu camu) (Experimental): Patients receive nivolumab IV over 30 minutes on day, ipilimumab IV over 30 minutes on day 1, and camu camu PO QD continuously with each cycle. Cycles repeat every 3 weeks for cycles 1-4. Beginning cycle 5, patients receive nivolumab over 30 minutes on day 1, and camu camu PO QD of each cycle. Cycles repeat every 4 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo blood and stool sample collection and undergo CT and/or bone scan and/or MRI on trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Biological: Ipilimumab; Procedure: Magnetic Resonance Imaging; Drug: Myrciaria dubia Prebiotic Supplement; Biological: Nivolumab

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood and stool sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; Ipilimumab Biosimilar CS1002; MDX-010; MDX-CTLA4; Yervoy
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Drug: Myrciaria dubia Prebiotic Supplement — Given PO
  Other Names: Camu Camu Prebiotic; Camu-camu Prebiotic; Myrciaria dubia based Prebiotic; Myrciaria dubia Supplement
  Arms: Arm 2 (nivolumab, ipilimumab, camu camu)
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; CMAB819; MDX-1106; NIVO; Nivolumab Biosimilar CMAB819; ONO-4538; Opdivo

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of camu camu when used in combination with nivolumab and ipilimumab in treating patients with kidney cancer that has spread to other places in the body. A monoclonal antibody is a type of protein that can bind to certain targets in the body, such as molecules that cause the body to make an immune response (antigens). Immunotherapy with monoclonal antibodies, such as nivolumab and ipilimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Camu camu is a prebiotic that may have a beneficial effect on the immune system. Giving camu camu in combination with nivolumab and ipilimumab may kill more tumor cells than nivolumab and ipilimumab alone in patients with metastatic kidney cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the effect of camu camu in combination with nivolumab/ipilimumab on Ruminococcus abundance in stool samples of patients with metastatic renal cell carcinoma (mRCC).

SECONDARY OBJECTIVES:

I. To evaluate the effect of camu camu on the clinical efficacy of the nivolumab/ipilimumab combination.

II. To determine the effect of camu camu on systemic immunodulation of the nivolumab/ipilimumab combination in patients with mRCC.

III. To describe the toxicity and safety profile of the use of camu camu in combination with nivolumab/ipilimumab.

IV. To determine the effect of camu camu on gut microbiome diversity and function.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM 1: Patients receive nivolumab intravenously (IV) over 30 minutes on day 1 and ipilimumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 3 weeks for cycles 1-4. Beginning cycle 5, patients receive nivolumab over 30 minutes on day 1 of each cycle. Cycles repeat every 4 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo blood and stool sample collection and undergo computed tomography (CT) and/or bone scan and/or magnetic resonance imaging (MRI) on trial.

ARM 2: Patients receive nivolumab IV over 30 minutes on day, ipilimumab IV over 30 minutes on day 1, and camu camu orally (PO) once a day (QD) continuously with each cycle. Cycles repeat every 3 weeks for cycles 1-4. Beginning cycle 5, patients receive nivolumab over 30 minutes on day 1, and camu camu PO QD of each cycle. Cycles repeat every 4 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo blood and stool sample collection and undergo CT and/or bone scan and/or MRI on trial.

After completion of study treatment, patients are followed up every 12 weeks until time of death or formal withdrawal from the study, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide informed consent for the trial
* Histological confirmation of renal cell carcinoma (RCC) with a clear-cell or sarcomatoid component
* Advanced (not amenable to curative surgery or radiation therapy) or metastatic (American Joint Committee on Cancer [AJCC] 8 stage IV) RCC
* Intermediate or poor risk disease by International Metastatic Renal Cell Carcinoma Database Consortium Criteria (IMDC) classification
* No prior systemic therapy for RCC with the following exception:

  * One prior adjuvant or neoadjuvant therapy for completely resectable RCC if such therapy did not include an agent that targets PD-1 or PD-L1 and if recurrence occurred at least 6 months after the last dose of adjuvant or neoadjuvant therapy
* Eastern Cooperative Oncology Group (ECOG) performance status < 2
* Measurable disease as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Males and females, ages >= 18
* Any ethnicity or race
* Adequate renal function defined as calculated creatinine clearance >= 30 milliliters per minute (mL/min) per the Cockcroft and Gault formula or Serum creatinine < 1.5 x upper limit of normal (ULN)
* Adequate liver function defined by aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 3 x ULN (< 5 x ULN if liver metastases are present), and total bilirubin < 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin up to 3.0 mg/dL)
* White blood cells (WBC) > 2,000/mm^3
* Neutrophils > 1,500/mm^3
* Platelets > 100,000/mm^3

Exclusion Criteria:

* Presence of untreated brain metastases. Patients with treated brain metastases must be stable for 4 weeks after completion of treatment and have documented stability on pre-study imaging. Patients must have no clinical symptoms from brain metastases and have no requirement for systemic corticosteroids amounting to > 10 mg/day of prednisone or its equivalent for at least 2 weeks prior to first dose of study drug. Patients with known leptomeningeal metastases are excluded, even if treated
* Favorable risk disease by IMDC classification
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways
* Any active or recent history of a known or suspected autoimmune disease or recent history of a syndrome that required systemic corticosteroids (> 10 mg daily prednisone equivalent) or immunosuppressive medications except for syndromes which would not be expected to recur in the absence of an external trigger. Subjects with vitiligo or type I diabetes mellitus or residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement are permitted to enroll
* Active interstitial lung disease (ILD)/pneumonitis or history of ILD/pneumonitis requiring treatment with systemic steroids
* Baseline pulse oximetry less than 92% "on room air"
* Current use, or intent to use probiotics, prebiotics, yogurt, bacterial fortified foods and other natural supplements =< 2 week prior to treatment initiation and during the period of treatment
* Any condition requiring systemic treatment with corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days prior to first dose of study drug. Inhaled steroids and adrenal replacement steroid doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
* Uncontrolled adrenal insufficiency
* Known medical condition (e.g., a condition associated with diarrhea or acute diverticulitis) that, in the investigator's opinion, would increase the risk associated with study participation or study drug administration or interfere with the interpretation of safety results
* Not recovered to =< Grade 1 toxicities related to any prior therapy before administration of study drug
* Women who are pregnant or breastfeeding
* History of myocarditis or congestive heart failure (as defined by New York Heart Association Functional Classification III or IV), as well as unstable angina, serious uncontrolled cardiac arrhythmia, uncontrolled infection, or myocardial infarction 6 months prior to study entry
* WBC < 2,000/mm^3
* Neutrophils < 1,500/mm^3
* Platelets < 100,000/mm^3
* AST or ALT > 3 x ULN (> 5 x ULN if liver metastases are present)
* Total bilirubin > 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin 3.0 mg/dL)
* Calculated creatinine clearance <30 millimeters per minute (mL/min) per the Cockcroft and Gault formula or serum creatinine > 1.5 x upper limit of normal (ULN)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-06 (Actual); Primary Completion 2026-03-14 (Estimated); Study Completion 2026-03-14 (Estimated)

PRIMARY OUTCOMES:
Abundance of ruminococcus in the stool | From baseline to week 12 of therapy
  Using a two-group t-test with a one-sided type I error of 0.05.

SECONDARY OUTCOMES:
Best overall response | Every 12 weeks for up to 3 years
  Response and progression will be evaluated in this study using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Will be examined using Fisher's exact test.
Progression-free survival (PFS) | Time from enrollment to progression date or date of death, whichever occurs first (Each cycle is 4 weeks)
  PFS, assessed as the duration of time from enrollment to progression, with camu camu in combination with nivolumab/ipilimumab vs nivolumab/ipilimumab alone. The difference in progression-free survival across the two groups will be explored graphically using Kaplan-Meier survival plots. Median progression-free survival time for each of the two arms will be reported and Cox Proportional Hazards model will be used to estimate the hazard ratio and its confidence interval.
Incidence of adverse events | Up to 30 days post-last dose of protocol therapy
  Will perform statistical analysis to compare the rates of all grade and grade >= 3 (per Common Terminology Criteria for Adverse Events version 5) treatment related adverse events between nivolumab/ipilimumab and nivolumab/ipilimumab with camu camu arms.

CONTACTS AND LOCATIONS:
Overall Officials: Sumanta K Pal, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States